CLINICAL TRIAL: NCT03043833
Title: Improving Access to Treatment for Anxiety and Depression Among French Canadians Using an Internet-Delivered Cognitive Behavior Therapy: A Randomized Controlled Trial
Brief Title: Internet-Delivered Cognitive Behavior Therapy for Anxiety and Depression Amongst French Canadians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universite de Moncton (Other)
Collaborators: Macquarie University, Australia (Other)
Responsible Party: Principal Investigator, France Talbot, Associate Professor, Universite de Moncton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: File 1516-077
Record Dates: First submitted 2017-01-30; First posted 2017-02-06 (Estimated); Last update posted 2018-05-01 (Actual); Status verified 2018-04

CONDITIONS: Major Depression; Anxiety Disorders
MeSH Terms: conditions — Depressive Disorder, Major; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wellbeing Course (Experimental): Will receive the French-Canadian version of the Wellbeing Course consisting of five lessons based on cognitive behavior therapy delivered through the Internet over eight weeks.
  Interventions: Behavioral: The Wellbeing Course
- Waitlist-control (No Intervention): The Waitlist Control Group will receive the French-Canadian version of the Wellbeing Course once the treatment group will have completed treatment.

INTERVENTIONS:
Behavioral: The Wellbeing Course — The Wellbeing Course (Titov et al., 2011) includes five online lessons:
  * Lesson 1 presents information on the prevalence of anxiety disorders and depression as well as on how they may interfere with life goals. This lesson also discusses how cognitive, behavioral and physical symptoms can contribute to poor emotional health.
  * Lesson 2 presents different strategies to generate realistic cognitions.
  * Lesson 3 describes strategies for physical de-arousal and for re-engaging in reinforcing activities.
  * Lesson 4 describes avoidance and safety behaviors in relation with anxiety and depression along with graded exposure.
  * Lesson 5 is about problem solving, relapse prevention and staying well.
  For each lesson, a "Do It Yourself" guide is included as well vignettes and additional material.
  Arms: Wellbeing Course

SUMMARY:
This study represents Phase II of a research program involving an international collaboration with Macquarie University (Sydney, Australia) to implement an Internet-based cognitive behavior therapy for the treatment of anxiety and depression in French-speaking Canadians from the Atlantic Provinces.

The primary objective is to establish the clinical efficacy of a French-Canadian self-guided format version of the Wellbeing Course by conducting a randomized-control trial where an experimental group will be compared to a waitlist control group. A secondary objective is to demonstrate the course's acceptability through participants' satisfaction with the course.

ELIGIBILITY:
Inclusion Criteria:

* Residing in New-Brunswick, Nova-Scotia, Prince Edward Island, or Newfound land & Labrador
* Having identified French as the first official language spoken and having good reading comprehension in French.
* Reliable Internet access
* Clinically significant levels of depression or anxiety reflected by significant scores on the following measures: PHQ-9 > 9, GAD-7 >7, Penn Stage Worry Questionnaire ≥ 45, Social Phobia Inventory ≥ 19, Panic and Agoraphobia Scale ≥ 19, or by answering yes to the question "Is anxiety or low mood a problem for you"
* Not currently participating in cognitive-behavioral therapy
* No changes in medication for 4 weeks prior to the study, nor any changes in medication for the next 2 months
* Willing to disclose personal information

Exclusion Criteria:

* Presence of psychotic symptoms
* Presence of severe depression as indicated by scores ≥ 23 on the PHQ-9, or a score > 2 on item 9 of the PHQ-9

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-01-30 (Actual); Study Completion 2018-03-30 (Actual)

PRIMARY OUTCOMES:
Changes in depression as assessed by the Patient Health Questionnaire-9 (PHQ-9) | Pretest, posttest (week 8), 3-month follow-up
  Symptoms of depression
Changes in anxiety as assessed by the Generalized Anxiety Disorder-7 (GAD-7) | Pretest, posttest (week 8), 3-month follow-up
  Symptoms of anxiety

SECONDARY OUTCOMES:
Changes in life satisfaction as assessed by the Satisfaction with Life Scale (SWLS) | Pretest, posttest (week 8), 3-month follow-up
  Life satisfaction as assessed by the SWLS (Diener et al.,1995)
Changes in health as assessed by the Short-Form Health Survey | Pretest (week 1), posttest (week 8), 3-month follow-up
  Physical and mental health as assessed by the Short-Form Health Survey (SF-12; Ware et al., 1998)
Changes in personality as assessed by the Self-administered Standardised Assessment of Personality - Abbreviated Scale | Pretest (week 1), posttest (week 8), 3-month follow-up
  Pathological personality traits as assessed by the Self-administered Standardised Assessment of Personality - Abbreviated Scale (SAPAS)
Changes in anxiety as assessed by the Penn State Worry Questionnaire (PSWQ) | Pretest (week 1), posttest (week 8), 3-month follow-up
  Symptoms of worry
Changes in social anxiety as assessed by the Social Phobia Inventory (SPIN) | Pretest (week 1), posttest (week 8), 3-month follow-up
  Symptoms of social anxiety symptoms
Changes in panic and agoraphobia as assessed by the Panic and Agoraphobia Scale (PAS) | Pretest (week 1), posttest (week 8), 3-month follow-up
  frequency and intensity of panic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: France Talbot, Ph.D., Study Director — Université de Moncton
Locations (1):
- Université de Moncton - Adult Clinical Psychology Laboratory, Moncton, New Brunswick, Canada

IPD SHARING:
Plan to Share IPD: Undecided
There is currently in place a memorandum of understanding with Macquarie University, our collaborators. This agreement allows for the sharing of data once personally identifiable information has been removed.